CLINICAL TRIAL: NCT00257179
Title: The Serum Tissue Factor Level in Lung Cancer Patients as a Prognostic Factor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700609
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2005-06

CONDITIONS: Lung Cancer
Keywords: Tissue factor; Lung cancer; Tissue factor protein inhibitor; Factor VII; Factor X
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
This study uses serum tissue factor and tissue factor inhibitor and factor VII to monitor the pre-coagulation status in lung cancer patients and to correlate the pre-coagulation status with clinical staging and prognosis.

DETAILED DESCRIPTION:
The staging of lung cancer was according to tumor size, involvement of lymph node and metastatic status. But there is a different prognosis in cancer patients of the same stage. The coagulation status of cancer patients was considered as an important possible prognostic factor. So in this study, we want to evaluate patients' coagulation status and find the relation of coagulation status and cancer status.

We thus propose a prospective study using coagulation factors in order to search for the relationship between cancer stage and pre-coagulation status in Taiwanese lung cancer patients. We will also evaluate the potential use of tissue factor as a prognosis predictor in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly-diagnosed lung cancer
* Serum from cancer-free healthy volunteers

Exclusion Criteria:

* Chronic renal failure or end-stage renal disease [ESRD] (creatinine [Cr] > 2 )
* Hyperlipidemia on statin therapy
* Acute myocardial infarction
* Tapal or Plavix use
* Active thromboembolic event
* Severe liver disease (> child B)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jen Yu, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan